CLINICAL TRIAL: NCT05512104
Title: Clinical Characters and Outcome of Acute Myeloid Leukemia Patients on Correlation to CD200 and CD56 Expression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Gamal Mohamed Abd Elaal, Assistant lecturer, Assiut University
Other Study IDs: CD200 and CD56 in AML
Record Dates: First submitted 2022-08-16; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bone marrow aspirate and biopsy — fiow cytometry of bone marrow aspirate

SUMMARY:
estimation of the clinical characters and out come of adult acute myeloid leukemia patients

• correlation of the estimated clinical characters and outcome to the expression of CD200

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a clonal malignant disease of the hematopoietic tissue. The diversity of the clinical, the hematological and the genetic features among patients with AML has been recognized. Considerable progresses in defining new diagnostic and prognostic markers have been applied in AML treatment. The detection of specific molecules in the leukemic cells has special relevance and is mandatory for the identification of certain subtypes of myeloid neoplasms (Arber

* CD200 is a trans-membrane cell surface glycoprotein belonging to the type1 immunoglobulin super family (Wright , ). Expression of CD200 is normally seen in some population of T and B-lymphocytes, neurons and endothelial cells (Wright). CD200 induces immunosuppression through engagement with CD200R, a cell-surface receptor homolog, which is expressed on leukocytes of myeloid lineage, including mast-cells, macrophages, basophils, dendritic cells as well as certain T-cell populations. CD200, which is frequently over expressed in AML blasts and is associated with a worse outcome. It has the potential to induce the formation of CD4+ CD25+ FoxP3+ regulatory T cells (Tregs), a subset of immunosuppressive T cells that are linked with a poor prognosis in AML (Coles ). Abstract Background: Acute myeloid leukemia (AML) escape from immunosurveillance by immunosuppression. CD200 and CD56 expression represented an independent prognostic factor in many hematological malignancies but its importance in AML patients remains to be identified. Methods: CD200 and CD56 expression were assessed in the bone marrow blasts for Fifty-two (51) newly diagnosed AML by flowcytometry before start of therapy. Conclusions: CD200 and CD56 positive expression by myeloblasts at diagnosis denote poor prognostic indicator and correlated with poor cytogenetic findings. CD200 could be used as therapeutic target in AML. Keywords: CD200- CD56- AML- Prognosis RESEARCH ARTICLE Clinical Significance of CD200 and CD56 Expression in Patients with Acute Myeloid Leukemia, Leukemic cells express leukemia-associated antigen, MHC, co stimulatory molecules and ligands for natural killer (NK) cells activating receptors, therefore leukemic cells are susceptible to be attacked by T and NK cells (el-Shami ). CD56 antigen, a 200-220 kDa cell surface glycoprotein, identified as an isoform of the neural adhesion molecules (NCAM) (Gattenlöhner ). CD56 firstly described as NK cell and then found in several hematopoietic malignancies including AML (Yoshida ). CD56 was associated with poor prognosis in patients with acute myeloid leukemia (Alegretti ). We herein, study the expression level of CD200 and CD56 in de-novo acute myeloid leukemia patients to estimate the prognostic value of their positive expressions individually in AML cases

ELIGIBILITY:
Inclusion Criteria:

1. newly diagnosed Adult patients with AML, were treated with 3+7 protocol consists of 3 days doxorubicin (45mg/m2 ) and 7 days cytarabine (100-200 mg/m2 IV continuous infusion over 24 hours

   Exclusion Criteria:
   * 1-Promyelocytic leukemia (M3)
2. Secondary acute myeloid leukemia
3. aml patients above the age of 60 yrs
4. aml patients with end organ failure
5. patient not candidate for (3+7)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: newly diagnosed Adult patients with AML, were treated with 3+7 protocol consists of 3 days doxorubicin (45mg/m2 ) and 7 days cytarabine (100-200 mg/m2 IV continuous infusion over 24 hours
Sampling Method: Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Prognosis of Acute Myeloid Leukemia Patients on Correlation to CD200 and CD56 Expression | 1 year
  Prognostic value of CD200 and CD56 in acute myeloid leukemia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Damiani D, Tiribelli M, Raspadori D, Sirianni S, Meneghel A, Cavalllin M, Michelutti A, Toffoletti E, Geromin A, Simeone E, Bocchia M, Fanin R. Clinical impact of CD200 expression in patients with acute myeloid leukemia and correlation with other molecular prognostic factors. Oncotarget. 2015 Oct 6;6(30):30212-21. doi: 10.18632/oncotarget.4901. PMID 26338961